CLINICAL TRIAL: NCT07146958
Title: Voluntary Intake of Seed Enhanced Lunch Foods
Brief Title: Soup and Bread Recipe Impacts on Ingestive Behavior
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Janet Novotny, Research Physiologist, USDA Beltsville Human Nutrition Research Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HS70 - Soup Meal Liking Study
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Obesity &Amp; Overweight
Keywords: chia seeds; satiety; weight management
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: This study will be a randomized crossover with three treatment periods. Subjects (n=24, approximately equal number of men and women) will be randomly assigned to a treatment sequence.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Lunch Meal (Placebo Comparator): A lunch meal will be provided that is comprised of soup and bread. These items will be made from standard recipes. This arm will be a placebo comparator to meals made with chia seeds or help seeds, which may provide extra satiety.
  Interventions: Other: Placebo
- Chia Enriched Lunch Meal (Experimental): A lunch meal will be provided that is comprised of soup and bread. These items will be made from standard recipes that have been enhanced with chia seeds, which may provide extra satiety compared to the standard recipes in the placebo arm.
  Interventions: Other: Chia seeds
- Hemp Enriched Lunch Meal (Experimental): A lunch meal will be provided that is comprised of soup and bread. These items will be made from standard recipes that have been enhanced with hemp seeds, which may provide extra satiety compared to the standard recipes in the placebo arm.
  Interventions: Other: Hemp seeds

INTERVENTIONS:
Other: Chia seeds — Chia seeds will be added to soup and bread recipes.
  Arms: Chia Enriched Lunch Meal
Other: Hemp seeds — Hemp seeds will be added to soup and bread recipes.
  Arms: Hemp Enriched Lunch Meal
Other: Placebo — The placebo will be food items that are not enriched with the intervention products.
  Arms: Control Lunch Meal

SUMMARY:
The goal of the study is to determine the likability of seeds incorporated into lunch foods. The study will provide a better understanding of ways to make recipe alterations that may promote health and fullness.

DETAILED DESCRIPTION:
The objective of this study is to investigate the likability and potential satisfying effects of seed-enhanced foods. Seed consumption, owing to its high nutritional and functional characteristics, has become popular in recent years. Chia seeds, tiny edible seeds also known as Salvia hispanica L., are derived from a plant of the Lamiaceae family that grows in arid or semiarid climates. Hemp seeds are derived from the hemp plant Cannabis sativa. Although these seeds may seem different in appearance and taste, they share many similarities regarding their nutritional/health benefits. These seeds are a rich source of essential fatty acids (omega-3 and omega-6) and antioxidants. In addition, both chia and hemp seeds are sources of plant-based protein. Seeds also contain dietary fiber, which is essential to keep the digestive system healthy. The Dietary Guidelines for Americans recommend that adults consume 22-34 grams of fiber daily depending on age and sex. However, more than 90% of women and 97% of men do not meet the recommended fiber intake. Several studies in the past have shown the beneficial impact of supplementation with high-fiber foods exerting positive effects on appetite control and short-term satiety. Chia seeds are rich in soluble fiber that helps to lower cholesterol and delay starch digestion potentially impacting appetite and satiety. Various studies have reported the beneficial effects of chia seed consumption on cardiovascular disease, diabetes, and hypertension. Only a few studies have been conducted to investigate the satiating effects of chia or hemp seeds. These studies have mostly examined the influence of chia seed or hemp seeds as a mid-morning snack on short-term satiety and energy intake. No studies have examined how the use of chia or hemp seeds as a lunch meal ingredient could impact satiety. Therefore, the main objective of the present study is to investigate likability and potential satisfying effects of seed-enhanced foods.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Younger than 25 years
* Known (self-reported) allergy or adverse reaction to study foods
* Women who have given birth during the previous 12 months or who are pregnant/lactating or who plan to become pregnant over the upcoming 6 months (which will overlap with the study period)
* Presence of diabetes, diverticulitis (inflammation of the large intestine), colitis (inflammation of the colon), celiac disease, Crohn's disease, irritable bowel syndrome, gastrointestinal disease, pancreatic disease
* History of bariatric surgery or other weight control surgery
* Removal of a portion of the stomach or gastrointestinal tract
* Actively trying to gain or lose weight at the time of the study recruitment or planning to gain or lose weight during the study periods
* Diminished sense of taste and/or smell
* Anorexia Nervosa and/or Bulimia
* Smoking, vaping, or use of tobacco products in the past 3 months
* Suspected or known physiological/mechanical gastrointestinal (GI) obstruction
* Use of certain medications or supplements (prescription or over-the-counter) that may interfere with the study objectives
* Unable or unwilling to give informed consent or communicate with study staff
* Self-report of alcohol or substance abuse within the past 12 months and/or current treatment for these problems (long-term participation in Alcoholics Anonymous is not an exclusion)
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the study plan

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2025-11-05 (Estimated); Study Completion 2025-11-05 (Estimated)

PRIMARY OUTCOMES:
Lunch food intake | 30 minutes after the start of the intervention
  Mass of food eaten at lunch, weighed in grams
Feelings of hunger | 30 minutes post treatment
  Visual Analogue Scale assessment of hunger, assessed by participants placing a mark on a line, measured as millimeters across the line, with larger values meaning more hungry. To answer the question "How hungry do you feel?" one end of the line will be labeled "I am not hungry at all" and the other end of the line will be labeled "I have never been more hungry." This question is part of a validated ingestive behavior questionnaire.
Feelings of satisfaction | 30 minutes post intervention
  Visual analogue scale assessment of meal satisfaction, assessed by participants placing a mark on a line, measured as millimeters across the line, with larger values meaning more satisfied. To answer the question "How satisfied do you feel?" one end of the line will be labeled "I am completely empty" and the other end of the line will be labeled "I cannot eat another bite." This question is part of a validated ingestive behavior questionnaire.
Feelings of fullness | 30 minutes post intervention
  Visual analogue scale assessment of fullness, assessed by participants placing a mark on a line, measured as millimeters across the line, with larger values meaning more full. To answer the question "How full do you feel?" one end of the line will be labeled "Not at all full" and the other end of the line will be labeled "Totally full." This question is part of a validated ingestive behavior questionnaire.
Ability to consume more food | 30 minutes post intervention
  Visual analogue scale assessment of ability to consume more food, assessed by participants placing a mark on a line, measured as millimeters across the line, with larger values meaning more able to eat more food. To answer the question "How much do you think you can eat?" one end of the line will be labeled "Nothing at all" and the other end of the line will be labeled "A lot." This question is part of a validated ingestive behavior questionnaire.
Desire to eat something sweet | 30 minutes post intervention
  Visual analogue scale assessment of desire to consume something sweet, assessed by participants placing a mark on a line, measured as millimeters across the line, with larger values meaning more greater desire to eat something sweet. To answer the question "Would you like to eat something sweet?" one end of the line will be labeled "Yes, very much" and the other end of the line will be labeled "No, not at all." This question is part of a validated ingestive behavior questionnaire.
Desire to eat something salty | 30 minutes post intervention
  Visual analogue scale assessment of desire to consume something salty, assessed by participants placing a mark on a line, measured as millimeters across the line, with larger values meaning more greater desire to eat something salty. To answer the question "Would you like to eat something salty?" one end of the line will be labeled "Yes, very much" and the other end of the line will be labeled "No, not at all." This question is part of a validated ingestive behavior questionnaire.
Desire to eat something savory | 30 minutes post intervention
  Visual analogue scale assessment of desire to consume something savory, assessed by participants placing a mark on a line, measured as millimeters across the line, with larger values meaning more greater desire to eat something savory. To answer the question "Would you like to eat something savory?" one end of the line will be labeled "Yes, very much" and the other end of the line will be labeled "No, not at all." This question is part of a validated ingestive behavior questionnaire.
Desire to eat something fatty | 30 minutes post intervention
  Visual analogue scale assessment of desire to consume something fatty, assessed by participants placing a mark on a line, measured as millimeters across the line, with larger values meaning more greater desire to eat something fatty. To answer the question "Would you like to eat something fatty?" one end of the line will be labeled "Yes, very much" and the other end of the line will be labeled "No, not at all." This question is part of a validated ingestive behavior questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Janet Novotny, PhD, Principal Investigator — United States Department of Agriculture (USDA)
Locations (1):
- U.S. Department of Agriculture, Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Only de-identified information will be shared.